CLINICAL TRIAL: NCT00383682
Title: Randomized, Placebo-Controlled, Double-Blind Cross-Over Trial of Opioids Versus Mexiletine in the Treatment of Postamputation Pain
Brief Title: Efficacy of Opioids and Mexiletine for the Treatment of Postamputation Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P01HD033990 (NIH); Project 2, P01HD33990
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-09

CONDITIONS: Amputation; Chronic Pain
Keywords: postamputation pain; phantom pain; stump pain; neuroma pain; opioid; mexiletine
MeSH Terms: conditions — Chronic Pain; Phantom Limb | interventions — Morphine; Mexiletine

INTERVENTIONS:
Drug: morphine and mexiletine

SUMMARY:
Persistent pain occurs in 50-85 percent of patients who experience the amputation of an extremity. This study will compare the effectiveness of morphine and mexiletine to placebo in the treatment of postamputation pain.

It is hypothesized that the effects of opioids and mexiletine on behavior and mental functioning in patients with postamputation pain are unlikely to be significant barriers to the clinical use of the drugs.

DETAILED DESCRIPTION:
The long-term objective of this research is to develop better clinical strategies for alleviating pain resulting from amputation of extremities. Amputation is the most radical form of nerve injury. The two major types of postamputation painful sequela are phantom pain and stump pain. Phantom pain has been defined as painful sensation perceived in the missing body part, or portion thereof (Merskey and Bogduk,1994). Phantom pain is the most distressing, and often difficult to treat, chronic neuropathic pain syndrome that results from direct injury to the peripheral or central nervous system. Recent epidemiological studies indicate that 50-85% of patients experience persistent pain following amputations. This controlled clinical trial will examine the role of opioid analgesics and local anesthetics in the treatment of phantom and associated stump pain resulting from amputations. Specifically, our objectives are to answer the following questions:

1. Does therapy with opioids and mexiletine result in better management of postamputation pain than treatment with placebo? Using a randomized, blinded, crossover clinical trial, the effectiveness of therapy with the opioid, morphine, and the oral local anesthetic, mexiletine, will be compared with placebo in the management of phantom and associated stump pain following amputations. The effectiveness of the treatment regimens will be judged by improvements in: a) The intensity of ongoing, stimulus-independent pain using established pain intensity and pain relief scales, b) Stimulus-evoked pain using quantitative sensory tests, and c) Impairment of function using established measures.
2. What are the relative effects of opioids and mexiletine on affective and cognitive function in patients with amputated extremities? Using established tests of neuropsychological function, mood, and psychosocial and physical impairment, affective and cognitive changes associated with the opioid and mexiletine therapies will be quantified and compared with changes associated with placebo treatment. These studies will help determine if the effects of opioids and mexiletine on affect and cognition are likely to limit the usefulness of the medications in the treatment of pain following amputations.

ELIGIBILITY:
Inclusion Criteria:

Adults (18 years or older) of both sexes and all races with persistent phantom and or stump pain for 6 months or longer following an amputation will be eligible for enrollment in the study.

Exclusion Criteria:

1) age less than 18 or over 85 years, 2) history of allergic reaction to the study drugs, i.e., morphine and mexiletine, 3) cardiac conduction defects such as second degree or complete heart block, or a myocardial infarction in the last 3 months, 4) severe pulmonary disease, 5) current history of alcohol or substance abuse, 6) seizures, dementia or encephalopathy, 7) pregnancy and nursing mothers, 8) chronic hepatic disease or hepatic failure, 9) hematological disease associated with leukopenia and/or thrombocytopenia, and 10) other terminal illness with a life expectancy of less than 6 months. 11) Finally, to avoid a bias in patient selection, patients who failed to achieve clinically significant pain relief to a previous optimal trial with morphine and/or mexiletine will be excluded. An optimal trial will be defined as minimum of 3 week trial with either agent using a drug titration paradigm where the dose of the drugs were increased at intervals of one week or less.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1997-07; Study Completion 2003-04

PRIMARY OUTCOMES:
Pain intensity (0-10 numerical rating scale)

SECONDARY OUTCOMES:
Pain relief (0-100%)
Functional activity (Multidimensional Pain Inventory activity and interference subscales

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasa N Raja, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Wu CL, Agarwal S, Tella PK, Klick B, Clark MR, Haythornthwaite JA, Max MB, Raja SN. Morphine versus mexiletine for treatment of postamputation pain: a randomized, placebo-controlled, crossover trial. Anesthesiology. 2008 Aug;109(2):289-96. doi: 10.1097/ALN.0b013e31817f4523. PMID 18648238